CLINICAL TRIAL: NCT05399563
Title: Medico-legal Assessment of Sexual Violence and Pregnancy Related Allegations Among Females Presented to Women's Health Hospital -Assiut University
Brief Title: Medico-legal Assessment of Sexual Violence-Assiut University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Othman, Principal investigator in Forensic, Assiut University
Other Study IDs: a100
Record Dates: First submitted 2022-03-21; First posted 2022-06-01 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Attempted Rape of Female
Keywords: Obtain a detailed history and examination

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
* Medico legal assessment of sexual assaults allegations of females presented to hospital and any associated violence.
* Assessment of cases of pregnancy associated violence with other related complications that have both medical and legal implications.
* Knowing role of VAW Unit in compacting female abuse offering support and authentication of suspicious claims

DETAILED DESCRIPTION:
The data will be obtained after informed consents from cases. These cases will be then analyzed in terms of:

* Verifying legal procedures as careful reviewing of public prosecution order and associated victim's identification documents if present
* Obtain a detailed history including personal information as age, marital status' residence and education; incident circumstances like assault characteristics as numbers of assailants, relationship to the victim' place of assault' frequency of assault and the time lapse between examination and last assault, etc ; gynecologic and obstetric history.
* General examination that include proper documentation of all visible injuries all over the body (type' direction' location' shape) and local examination of genital or anal region and possibility of taking vaginal and anal swabs if possible.
* Re-examined victim after two weeks for exclude any venereal diseases and doing pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* All females above ≥ 12 years old with suspicious sexual violence or illegal pregnancy or criminal induction of abortion.

Exclusion Criteria:

* All females who will present to the women's health hospital above 12 years old for ordinary medical advice or treatment of gynecologic or obstetric complaints

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: As nature of a descriptive study design; All eligible cases of substance abuse admitted to Women Health Hospital and Safe Women's Unit belong to Assiut will be examined for inclusion and exclusion criteria. The cases will be included in the study in duration of one year (March 2022- February 2023).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-05-28 (Estimated); Study Completion 2023-05-28 (Estimated)

PRIMARY OUTCOMES:
Measure the prevalence of sexual violence problem among females | from 1-6-2022 to 28-5-2023
  These cases will be then analyzed in terms of Verifying legal procedures as careful reviewing of public prosecution order and associated victim's identification documents if present

IPD SHARING:
Plan to Share IPD: No